CLINICAL TRIAL: NCT03483532
Title: Study of the Crystallization Inhibition Capacity of the Uric Acid in Urine in a Group of Lithiasic Patients After Intake of a Food Supplement. PEv2
Brief Title: Study of the Crystallization Inhibition Capacity of the Uric Acid in Urine in a Group of Lithiasic Patients After Intake of a Food Supplement
Status: Completed | Type: Observational
Sponsor: Devicare S.L. (Industry)
Collaborators: Universidad de las Islas Baleares (Unknown)
Responsible Party: Sponsor
Other Study IDs: IB 3414/17
Record Dates: First submitted 2018-02-06; First posted 2018-03-30 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Lithiasis
Keywords: lithiasis; uric acid; crystallization
MeSH Terms: conditions — Lithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Biospecimen Retention: Samples Without DNA — Urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lit Control pH Up without cocoa extract: The nutritional exposure will consist in the intake of 1 capsule of the food supplement based on citrate and plant extract without cocoa extract dosed at the rate of one during breakfast and another during dinner, during a period of 14 days to a group of 30 patients.
  Interventions: Dietary Supplement: Lit Control pH Up
- Lit Control pH Up with dry cocoa extract: The nutritional exposure will consist in the intake of 1 capsule of the food supplement based on citrate and plant extract with cocoa extract dosed at the rate of one during breakfast and another during dinner, during a period of 14 days to a group of 30 patients.
  Interventions: Dietary Supplement: dry cocoa extract

INTERVENTIONS:
Dietary Supplement: Lit Control pH Up — dietary supplement based on citrate, saponins, magnesium, zinc and vitamin A
  Groups: Lit Control pH Up without cocoa extract
Dietary Supplement: dry cocoa extract — (Theobroma cacao, fruit), 2 capsules of 750 mg per individual, dosed at a rate of one during the breakfast and another during dinner.
  Groups: Lit Control pH Up with dry cocoa extract

SUMMARY:
Renal lithiasis affects a wide range of the population, ranging from 4 to 15% according to the population sample studied. Among all stones, it is estimated that uric stones account for between 10 and 15% of all cases and especially affects men over 50 years, while mixed lithiasis of calcium oxalate monohydrate and uric acid affects a 2.5% of all cases. Lithiasis generated by uric acid is a highly recurrent pathology, even repeating itself several times during the year, and is related to other pathologies such as diabetes and obesity. It is evident that the medical problem that lithiasis originates should not be treated only by eliminating the calculus formed, through the different surgical techniques available, but also that the alterations responsible for its formation should be modified and corrected. If these alterations are not modified, the risk of the genesis of new calculations persists.

The pharmacological treatments used until now to treat uric lithiasis are based on the powerful alkalinization of the urine (through the use of citrate or bicarbonate); These treatments tend to have a low rate of adherence and, taken long term, can cause the development of stones of another composition (eg, Phosphate), which are much more difficult to treat.

There are natural substances, such as theobromine (natural component of cocoa) that has been found to have the ability to inhibit the formation of uric acid crystals: this substance has been tested in laboratory experiments and therefore would be useful to prevent the formation of uric acid stones and / or mixed calcium oxalate monohydrate / uric acid stones. Theobromine corresponds to a phytocomponent alkaloid that is found in high concentrations in chocolate. The starting hypothesis of this study corresponds to the possible increase in the capacity of inhibition of the crystallization of uric acid by urine in subjects who have ingested food or food supplements containing cocoa or cocoa extract. Therefore, the relationship between the intake of a specific food supplement and the ability to inhibit the crystallization of uric acid by the urine will be studied. An increase in the ability to inhibit the crystallization of uric acid from urine would be useful to prevent the formation of uric acid crystals in urine, which are the origin of uric acid stones or mixed calcium oxalate monohydrate / acid uric.

Currently there is no information on the relationship between the ability to inhibit the crystallization of uric acid in the urine due to the intake of certain foods or food supplements and the concentration of theobromine in urine and urinary pH. The present study is carried out to evaluate the relationship between the intake of a specific food supplement and the ability to inhibit the crystallization of uric acid by urine, which would be useful to prevent the formation of uric acid stones and / or mixed calculations of calcium oxalate monohydrate / uric acid.

The study will be carried out in two stages. The first will consist in the intake of 1 capsule of a food supplement based on citrate and plant extract without cocoa extract, twice a day for 14 days. The second will consist in the intake of 1 capsule of a food supplement based on citrate and plant extract with cocoa extract, twice a day for 14 days. Before the start of the study a blood sample will be obtained and on the last day of each stage, the patient will be asked to collect the 24-hour urine and another 2-hour morning urine sample. Between each stage will be a period of 7 days without receiving any food supplement.

During the study there will be no risk due to the tests that will be performed, since they are among those performed in routine clinical practice. Regarding the possible risks associated with the intake of food supplement, to minimize them, any patient with chocolate or theobromine allergy, pregnant or lactating women and patients with insufficiency are excluded from the study participation. chronic kidney The daily amount of theobromine ingested as cocoa extract is similar to a quantity of dark chocolate between 11-25 g. This consumption of chocolate can be considered normal within a diet. In fact a piece of 50 g of dark chocolate contains between 237 and 519 mg of theobromine and daily many people consume more of this amount without presenting side effects to be a food.

DETAILED DESCRIPTION:
Background Urolithiasis is a pathology known since antiquity although they are not known totally the causes of the formation of all the different types of calculus existing As a consequence of this, only in some cases has it been possible to develop an efficient treatment. Renal lithiasis affects a wide range of the population, varying from 4 to 15% according to the population sample studied. It is important to highlight the high morbidity associated with this pathology, since between 10 and 15% of cases require surgical treatment and between 20 and 30% it requires hospitalization. Among all lithiasis, it is estimated that uric lithiasis accounts for between 10 and 15% of all cases and especially affects men over 50 years old, while mixed lithiasis of calcium oxalate monohydrate and uric acid affects 2.5% of all the cases. Lithiasis generated by uric acid are a highly pathology recurrent, even repeating several times during the year, and is related with other pathologies such as diabetes and obesity. This implies a high cost estimated in billions of euros per year, especially for its incidence in medical emergencies. It should be noted that between 50 and 70% of people who do not receive treatment or do not change their nutritional habits develop new calculus in a period of time less than 5 years. Is a contracted fact that the type and characteristics of the feed will determine the functioning of the acid-base metabolism and the characteristics of the urine as it can be its pH, the greater or lesser concentration of substances, as well as a set of characteristics that can determine the crystallization capacity of the different substances contained in it such as uric acid. It is evident that the medical problem that lithiasis originates should not be treated so only eliminating the same one, by means of the different surgical techniques available, but also the alterations responsible for its use must be modified and corrected training. If these alterations are not modified, the risk of genesis of new calculus persists. The pharmacological treatments used so far for treat uric lithiasis are based on the powerful alkalinization of urine (by using of citrate or bicarbonate) increasing the urinary pH to avoid crystallization of the uric acid and the formation of new kidney stones. These treatments can present a long-term problem and as a consequence there is a low- 2 - percentage of adherence to the treatment of uric acid stones. These long-term treatments can increase urinary pH above 6 units and end up causing a different type of renal lithiasis, the phosphatic, a lot more difficult to treat, by increasing the possibility of total calcification of the kidney that it implies. Therefore, it is evident that new alternatives should be sought in substances of food source that could facilitate the dietary treatments of said pathology.

There are currently citrate-based food supplements on the market plant extracts that contribute to the normal functioning of the metabolism acid-base of the organism alkalizing the urine (for example Lit control pH up). But there are also other approaches to the problem of lithiasis based on avoiding or decreasing the crystallization capacity of urine developed by the Renal Lithiasis Research Laboratory of the University of the Illes Balears. These approaches consist in looking for inhibitors of the crystallization of natural origin A crystallization inhibitor corresponds to a substance that is able to prevent, delay or hinder the crystallization of insoluble compounds. This approach was already started with the work of Bliznakov in 1965, showing that certain molecules were able to slow down the growth rate crystalline nature of certain substances as a result of their adsorption (binding) on growth surfaces and the corresponding alterations that this caused. During this time Vermeulen et al., Fleisch et al. and Howard and cols showed that a series of substances present in the urine, including pyrophosphate, were capable to prevent the crystallization of the calcium salts. These ideas too were later developed by the Lithiasis Research Laboratory Renal observing that said inhibitory capacity of the crystallization of calcium salts It was also made by phytate, a substance that is present in all unrefined seeds (legumes, cereals, nuts, ...). This process led to the search for natural substances that presented said ability to inhibit, not on the crystallization of calcium salts but on the crystallization of uric acid. Among numerous substances used in the tests In vitro it was observed that theobromine, natural component of cocoa produces said effect concentrations similar to those produced after the usual chocolate intake. In Europe chocolate intake is approximately between 6 and 12 kg per person and year. For this reason, it is intended to reduce the inhibition capacity of the uric acid from the urine by an in vitro test after the intake of a supplement determined food For this purpose, urine samples from patients will be used volunteers who will supply to the Renal Lithiasis Research Laboratory assigned to the IUNICS (University of the Balearic Islands) before and after the intake of- 3 - a certain food supplement food for a time settled down.

Justification The Renal Lithiasis Research Laboratory since 1998 has as one of its its purpose is to study the relationship between the characteristics of urine and the different types of existing lithiasis. As we have indicated one of the lithiases with a large incidence is lithiasis of uric acid or calcium oxalate monohydrate / uric acid. Currently, the relationship between the ability to inhibit crystallization of uric acid from a urine after ingestion of certain food Complements.

Urine is a product of blood filtration that reflects its composition, including water and low molecular weight molecules such as salts, vitamins, minerals, etc. accordingly the intake of certain foods, such as the chocolate, cocoa or an extract thereof, will be reflected in an increase in urinary excretion of theobromine, an inhibitor of the crystallization of uric acid.

Due to this, the modification of the crystallization capacity of uric acid in the urine should be clearly reflected. Naturally, apart from this main variable, urine must be determined in series of secondary variables such as urinary pH, concentration of Theobromine and all other important urinary parameters in the pathology lithiasic.

Main objective and secondary objectives Currently, the relationship between the ability to inhibit crystallization of uric acid by urine due to the intake of certain food or food supplements and theobromine concentration and pH urinary. Therefore, the main objective is to evaluate the inhibition capacity of the crystallization of uric acid by urine in patients diagnosed with uric lithiasis or calcium oxalate monohydrate / uric acid, after ingestion of a food supplement with cocoa extract. This would allow to use the capacity of inhibition of the crystallization of uric acid by urine, as a possible indicator of the prevention of uric lithiasis or calcium oxalate monohydrate / acid uric due to the effect of food.

Hypothesis The starting hypothesis of this study corresponds to the possible increase in ability to inhibit the crystallization of uric acid by urine from subjects who have eaten foods that contain cocoa or cocoa extract. Thus the relationship between the intake of a specific complement will be studied nutritional status and the ability to inhibit the crystallization of uric acid by the urine. An increase in the ability to inhibit the crystallization of uric acid of urine would be useful to prevent the crystallization of uric acid, which is the origin of uric acid stones or mixed calcium oxalate monohydrate / acid uric stones.

Work design and methodology Study group The inhibitory capacity of the uric acid crystallization of urine will be studied in two groups of patients who will be proposed to take the food supplement based on citrate and plant extracts and the citrate-based food supplement and extracts of plants with cocoa extract during a period of 14 days. To these groups will be supplied with the food supplement that they should consume during the period of 14 days along with your usual diet.

Dietary intervention The food supplement to be consumed will be Lit Control pH Up without dry extract of ginseng (Panax ginseng, root) and the same Lit Control pH Up with dry cocoa extract (Theobroma cacao, fruit) that correspond to the capsules with cocoa extract. The dose will be 2 capsules of 750 mg per individual, dosed at a rate of one during the breakfast and another during dinner. Each participant will be provided with free the necessary number of nutritional capsules of the nutritional intervention.

Composition of nutritional supplements of the nutritional intervention (capsule of 750 mg of weight)

* Lit control pH up (with dry cocoa extract): Potassium citrate, citrate magnesium, dry extract of cocoa (Theobroma cacao, 60 mg of theobromine), maltodextrin (bulking agent), silicon dioxide (anticaking), magnesium stearate (fluidizing), zinc gluconate, vitamin A. Coverage: gelatin, titanium dioxide (opacifier), rust yellow iron (dye), indigotine-FD & C Blue2 (dye). CN: 172249.2. Weight capsule 750 mg
* Lit control pH up (without dry cocoa extract): Potassium citrate, citrate magnesium, maltodextrin (bulking agent), silicon dioxide (anticaking), magnesium stearate (fluidizing), zinc gluconate, vitamin A. Coverage: gelatin, titanium dioxide (opacifier), rust yellow iron (dye), indigotine-FD & C Blue2 (dye). Weight 750 mg capsule Absence of adverse / secondary effects of the food supplement Theobromine corresponds to a phytocomponent alkaloid found in high concentrations in chocolate, in fact a piece of 50 g of chocolate black contains between 237 and 519 mg of theobromine and daily many people consumes more than this amount without presenting side effects as it is a food. It is evident that the daily amount of theobromine ingested as an extract of cocoa would roughly correspond to a quantity of chocolate located between about 11-25 g, amount of consumption that can be considered normal on a diet. In a paper by Birkett et al (1985) where 200 mg of theobromine was ingested orally Three times a day, no clinical symptoms or pharmacological activity were observed. Nor the intake of theobromine as sweet chocolate at a dose of 6 mg / kg · day (for a person of 70 kg correspond to 420 mg / day of theobromine) causes effects Clinical trials in human subjects (Shively et al., 1985). There are different studies that determine the effect of theobromine on mood and use amounts of theobromine located around 700 mg / day as described in Mitchell et al. (2011). Finally, in a study that compared the ingestion of theobromine at doses 250 mg compared to placebo, there were no significant differences in the increased heart rate neither in systolic or diastolic blood pressure (Baggott et al., 2013).The WHO report (1991) describes that the ingestion of high doses of theobromine in human daily intakes of chocolate from 50-100 g of cocoa (0.8-1.5 g of theobromine) may be associated in some cases with sweating, trembling and pain of head This is a dose about eight times higher than that used in the intervention dietetics.

For all the exposed data it is evident that the theobromine existing in the extract of cacao that they will ingest in the dietetic intervention is far from any effect toxic. This nutritional dosage corresponds to a normal intake of Theobromine in the form of chocolate.

Main goal The present observational research project aims to evaluate the activity of a food supplement Lit Control pH Up without dry ginseng extract compared to another Lit Control pH Up with dry cocoa extract in lithiasic subjects normouricemic with uric acid lithiasis and / or COM / Ac. demonstrated uric acid, during a period of 14 days of intervention. The main variable of study will be the capacity of inhibition of the crystallization of uric acid in the first morning urine of 2 h.

Secondary objective Know the profile of the blood and urinary biochemical parameters of the patients recruited in the nutritional intervention.

Study design Non-randomized observational trial crossed and open to single blind. Definition of the study population: selection criteria

Subjects with uric lithiasis or urinary COM / Ac diagnosed, will be included in the study. not hyperuricemic, it is understood as such the existence of at least one episode previous with external elimination of the calculation by spontaneous expulsion, extracorporeal lithotripsy or other surgical techniques and subsequent analysis and identification of the same as well as the absence of demonstrable hyperuricemia from the data of:

* Clinical history, physical examination with TA control and explorations complementary
* Simple abdominal x-ray (urinary system)
* Biochemical and urinary analysis

Inclusion criteria:

The patient:

* You are over 18 and less than 75 years old
* You have presented a previous episode of objectifiable uric lithiasis
* Presents normouricemia
* Possesses the results of laboratory tests (biochemistry and urine)
* The patient agrees to participate and collaborate in the study

Exclusion criteria:

The patient presents:

* Active urinary infection
* Allergy to chocolate or theobromine
* Serum creatinine greater than 1.5 mg / dl
* Pregnancy, lactation period (women)
* Intestinal obstruction
* Hyperuricemia
* Treatment with diuretics
* Treatment with allopurinol or febuxostat.
* Congestive heart failure
* Other pharmacological treatments for the prevention of hyperuricemia
* Chronic renal failure Population sample of the intervention The number of patients will be 60 (see the justification for the number of patients in the section Study sample). This intervention will be carried out in a sample of patients with uric lithiasis or urinary COM / Ac uric acid, as it is a sample of patients available. This corresponds to a preliminary study and its use does not allows a direct extrapolation of the data obtained to the general population. This available sample will be described sufficiently to be able to make a cautious extrapolation to the population that could be represented by that sample. The studies with these population samples are the ones that are used to make specific studies on the same samples and to carry out studies experimental with few subjects as is this case.

Recruitment route The sample of voluntary patients will be recruited by the Urology Service of Hospital de Manacor among its patients who meet the inclusion criteria and not the exclusion criteria described above.

Observation period The investigator must recruit a minimum of 60 patients from observational form and with the data collected from the existing clinical histories, during a period of 36 months, considering the time required for the recruitment.

Description of the nutritional intervention Stage 1. The nutritional exposure will consist in the intake of 1 capsule of the food supplement based on citrate and plant extract without cocoa extract dosed at the rate of one during breakfast and another during dinner, during a period of 14 days to a group of 30 patients.

Stage 2. The nutritional exposure will consist in the intake of 1 capsule of the food supplement based on citrate and plant extract with cocoa extract dosed at the rate of one during breakfast and another during dinner, during a period of 14 days to a group of 30 patients.

After each stage, a week of bleaching will be carried out and the Initial assigned nutritional intervention. Each patient is assigned randomly from successive to Stage 1 or Stage 2.

Selection of the control group In this intervention there is no control group, the own The individual will be evaluated before and after the nutritional intervention.

Study sample. Predetermination of sample size The fact that it is a pilot study and carried out under conditions of clinical practice usual and have little information about the action of the complement food complicates the realization of the hypothesis. For what has not been done initial sample size calculation, because it is an observational pilot study Initial post-marketing modification of the urine characteristics of the patient. The choice of 60 subjects is decided in agreement with the researchers.

Subjects withdrawn due to intolerance will not be replaced and will be included in the analysis of data. Patients who leave the study due to any other circumstance, they must be replaced and will not be included in the statistical analysis. No relevant factors influence such as inclusion and exclusion criteria, since each patient serves as his own control. Variability is reduced, which is why you need a smaller sample size, in order to detect statistical difference between the intervention group and the control group. The cross study allows to evaluate the response to treatment in a short period of time, and the first intervention did not interferes with that of the second stage. The period of bleaching or "washing" (wash-out) between the two stages allows to avoid possible interferences between interventions of the first stage and the second.

Data collection notebook In research projects where the characteristics of samples are studied and that do not correspond to clinical trials of new drugs is not needed the CRF so it is not used in this research project (Law 14/2007, of July 3, of Biomedical Research). This study does not create personalized data file since only the urine sample is used will be anonymized by not using any personal data.

Process The study will involve for each patient the following operations not included in the usual clinical practice. Obtaining morning urine for 2 hours and collecting urine for 24 hours according to the instructions before each dietary intervention. Obtaining the 2-hour morning urine collection of 24-hour urine according to the instructions the last day of the dietetic intervention for each of the two study groups. The Patients will deposit their samples in the Urology Department of the Regional Hospital of Manacor to your usual doctor. The recruited patients will voluntarily cede to the Renal Lithiasis Research Laboratory of the UIB its urine samples for the realization of the test of the inhibition capacity of acid crystallization uric acid, the main variable of study and the determination of theobromine by high pressure liquid chromatography technique and annualized detection through an ultraviolet detector. The other biochemical determinations shall be carried out according to the protocols established in the usual clinical practice at the Hospital Comarcal of Manacor.

Study variables Sociodemographic variables

* Age: years (year of birth)
* Gender: male / female
* Weight / height and BMI Clinical variables The variables to analyze will be

  * Blood pressure
  * Intrinsic and extrinsic factors of the patient
  * Date of onset of symptoms
  * Symptoms and accompanying signs
  * Personal history
  * Previous treatments
  * Adverse effects attributable to nutritional intervention: Adverse effects they will be recorded when they appear in the clinical history or when in the clinical history there are clinical signs and symptoms that make it possible to define them as such.

Biochemical variables The study variables will be the following blood biochemical parameters and urinals that correspond to the standardized controls of lithiasic patients: 24-hour urine

* Creatinine
* Phosphate
* Uric acid
* Oxalate
* Citrate
* Calcium
* Magnesium

  2-hour urine
* Creatinine
* pH
* Ability to inhibit the crystallization of uric acid. Main variable of study Blood plasma
* Creatinine
* Phosphate
* Calcium
* Magnesium
* Potassium
* Uric acid The blood and urine analysis of 24 hours will be performed at the Hospital de Manacor (within usual clinical practice), the surplus will be destroyed according to the protocols established for the samples analyzed as in any other patient. The analytical carried out on the urine for 2 hours (which is the one that will be carried out in the Laboratory of research in renal lithiasis of the University of the Balearic Islands IUNICS), I do not know foresees that there are surpluses of urine samples. In case it exists, it will will be destroyed according to the protocols established for said samples by the Renal lithiasis research laboratory.

Schedule of activities

* Planned start corresponds to the second quarter of 2017 (conditioned final authorization CEIC).
* The planned completion corresponds to the third quarter of 2018. Statistic analysis A descriptive analysis of all the demographic and analytical data of the volunteers. The continuous quantitative variables will determine the average as measure of centralization while the variability will be defined by the deviation typical and the coefficient of variation. The statistical analysis of the variables will be carried out by means of the Student t test for paired samples for the determination of differences between the two sample means and for the construction of the interval of trust. The test checks whether the means of two samples distributed in a normal shape are the same.

ELIGIBILITY:
Inclusion Criteria:

* You are over 18 and less than 75 years old
* You have presented a previous episode of objectifiable uric lithiasis
* Presents normouricemia
* Possesses the results of laboratory tests (biochemistry and urine)
* The patient agrees to participate and collaborate in the study

Exclusion Criteria:

* Active urinary infection
* Allergy to chocolate or theobromine
* Serum creatinine greater than 1.5 mg / dl
* Pregnancy, lactation period (women)
* Intestinal obstruction
* Hyperuricemia
* Treatment with diuretics
* Treatment with allopurinol or febuxostat.
* Congestive heart failure
* Other pharmacological treatments for the prevention of hyperuricemia
* Chronic renal failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The number of patients will be 60 (see the justification for the number of patients in the section Study sample). This intervention will be carried out in a sample of patients with uric lithiasis or urinary COM / Ac uric acid, as it is a sample of patients available. This corresponds to a preliminary study and its use does not allows a direct extrapolation of the data obtained to the general population. This available sample will be described sufficiently to be able to make a cautious extrapolation to the population that could be represented by that sample. The studies with these population samples are the ones that are used to make specific studies on the same samples and to carry out studies experimental with few subjects as is this case.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Inhibition of the crystallization of uric acid | 12 hours
  Capacity of inhibition of the crystallization of uric acid in the first morning urine

SECONDARY OUTCOMES:
Uric Acid | 12 hours
  Uric Acid in Urine, measured in mg/L
Creatine | 12 hours
  Creatine in urin, measured in mg/L
Oxalate | 12 hours
  mg/L
Teobromine | 12 hours
  Teobromine in urine, measured in mg/L
Urine Volume | 12 hours
  Measured in ml
pH | 12 hours
  Urine ph

CONTACTS AND LOCATIONS:
Overall Officials: Fèlix Grases Freixedas, Principal Investigator — Universidad de las Islas Baleares; Yumaira Elena Hernández Martínez, Principal Investigator — Hospital de Manacor
Locations (1):
- Hospital de Manacor, Manacor, Balearic Islands, Spain